CLINICAL TRIAL: NCT04100278
Title: Effectiveness of Shared Care Diabetes Management in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Professor and Director, Department of Endocrinology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCDM-T2DM
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Diabetes Education and Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomization, parallel, controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional therapy group (No Intervention): All patients in this group will be given routine diabetes management, including lifestyle education, health guidance, monitoring blood sugar guidance and drug adjustment.
- Shared Care group (Active Comparator): The patients download the Shared Care mobile application and connect with the smart-glucometer Bg1 to upload blood glucose dairy in real time. With patient's informed consent, his or her data from each visit will be collected and recorded for analysis. After the patient returns home from the clinic, they can communicate through the APP with online diabetes educators. According to protocol, online diabetes educators answer patients' questions, give suggestions on patients' diet and summarize patients' issues to physicians, who provide high level supervision.
  Interventions: Behavioral: Shared Care diabetes management

INTERVENTIONS:
Behavioral: Shared Care diabetes management — After the inclusion visit, the patients will be randomized to Shared Care group or traditional therapy group. Compared to conventional diabetes education in the traditional therapy group, the Shared Care group provides patients with online services and continuous diabetes management and education through a mobile application. It also addresses that it is important for patients to meet regularly with diabetes multidisciplinary team for better results. The total observation period is 3 years for each patient. The visits will be done every 3 months.
  Arms: Shared Care group

SUMMARY:
This is a prospective, randomization, parallel, controlled study to evaluate the effectiveness of Shared Care diabetes management. Patients with T2DM involved in the Shared Care model pay regularly quarterly visit to a multidisciplinary team led by physician at outpatient clinic, and receive remote patient management and education after going home. After at least 3 years follow-up, patients' metabolic indexes including HbA1c, LDL-c, blood pressure, diabetes self-management behavior indexes and diabetes complications are evaluated.

The primary goal is to observe the HbA1c levels and the HbA1c achieving rate. The secondary goal is to assess the diabetes self-management behavior change for patients of the Shared Care multidisciplinary diabetes care model and to assess the effect of online diabetes self-management support for patients of the Shared Care multidisciplinary diabetes care model.

DETAILED DESCRIPTION:
With population aging and increasing prevalence of obesity in China, the number of patients with diabetes mellitus, healthcare expenditure and mortality related to DM are forecast to grow substantially. 114 million diabetic patients and 11.6% incidence rate of diabetes yield enormous chronic disease management pressure. China medical resources are not sufficient for the great diabetes epidemic (1-5) . The data from a multicenter, cross-sectional survey of outpatients conducted in 606 hospitals across China showed that the majority of patients with type 2 diabetes did not achieve the goal of HbA1c <7.0% (6). We are facing problems including inadequate patient education, unable to track the entire diabetic course, and the lack of effective patient engagement in-between clinic visits(1-5). Diabetes management and education can improve patients' quality of life, reduce incidence and mortality of diabetic complications and relieve the medical economy burden for the government. (7).

International guidelines published by American Diabetes Association and the National Institute and Health and Care Excellence in Hong Kong imply that a chronic disease service delivery model that incorporates continuous follow-ups, DSMES (diabetes self-management education and support) with a multidisciplinary team of health professionals to provide ongoing treatments, patient education, and scheduled health assessments for monitoring of disease control and complications has promoted internationally as a more holistic and cost-effective way to manage patients with diabetes(8-12) . To help health professionals to improve medical efficiency and help patients develop healthy lifestyle, we established Shared Care diabetes management model and believe that it can provide a solution.

Shared Care Model aims to empower patients with diabetes self-management education and supports (DSMES), achieve better health outcomes and delay incidence and mortality of diabetic complications. Compared with traditional diabetes outpatient settings, patients of Shared Care return to the hospital for regular follow-up every three months, and meet with a multidisciplinary team includes diabetes educators, nurses, dietitians and physical therapist led by the physician. The patients download the Shared Care mobile application during the outpatient service and connect with the smart-glucometer Bg1 to upload blood glucose dairy in real time. With patient's informed consent, his or her data from each visit will be collected and recorded for analysis.

The internet, IOT (internet of Things) and other information technology enables the Shared Care model to integrate outpatient and remote patient management, online and face-to-face medical services and provide patients with comprehensive health care. Our health care extended beyond the hospital. After the patient returns home from the clinic, they can communicate through the APP with online diabetes educators. The educators answer patients' questions, give suggestions on patients' diet and summarize patients' issues to physicians, who provide high level supervision. The model enables both patients and medical team for real-time data sharing, smart analysis and remote monitoring which significantly improve management efficiency and release medical resources for more patients.

The Shared Care program in our hospital was established since Jan. 2018. Until Jul. 2019, there are totally 1062 patients receiving continuous diabetes care which was provided by a multidisciplinary team. 82.8% patients are followed regularly every three months, the HbA1c achieving rate (<7%) is 69.5% after 1-year follow-up. Patient's self-management behavior improves one year after admission. The study is aim to discover the influencing factors that affect the HbA1c achieving rate and the efficiency and effect of the new model Shared Care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with T2DM
* Patients who have Informed and signed the consent form content
* Patients can be regularly followed (every 3 months) for at least 3 years

Exclusion Criteria:

* Patients with important organ failure or other severe diseases including infection, mentally disorder, heart failure or disseminated intravascular coagulation
* Patients with active or inactive malignant tumour, expectation of life less than 1 year
* Patients with communication disorders, cannot communicate and/or cooperate
* Females that are regnant, breast-feeding female, or conception plan in the recent year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c change | through study completion, an average of 3 year
  The change between baseline HbA1c and HbA1c 3 years after admission
Blood Pressure change | through study completion, an average of 3 year
  The change between baseline blood pressure and blood pressure 3 years after admission
LDL-c change | through study completion, an average of 3 year
  The change between baseline LDL-c and LDL-c 3 years after admission

SECONDARY OUTCOMES:
BMI change | through study completion, an average of 3 year
  The change between baseline BMI and BMI 3 years after admission, BMI is body mass index, weight and height will be combined to report BMI in kg/m^2
SDSCA(Summary of Diabetes Self Care Activities) score change | through study completion, an average of 3 year
  The change between baseline SDSCA score and SDSCA score 3 years after admission, SDSCA is scale Summary of Diabetes Self Care Activities (SDSCA), with 12 questions, each provide a minimum of 0 and maximum of 7 scores (7 indicates better self care action), total score 84
C-DMSES(Chinese Diabetes Management Self-Efficacy Scale) score change | through study completion, an average of 3 year
  The change between baseline C-DMSES and C-DMSES 3 years after admission. C-DMSES is Chinese Diabetes Management Self-Efficacy Scale. The scale measures the self-efficacy level of diabetes management. The C-DMSES has 20 questions, each question has a minimum score of 0 (indicates lowest self-efficacy), maximum score of 10(indicates highest self-efficacy). the scale has totally 200 scores.
A-DQOL(Amendment Diabetes Quality of Life scale) score change | through study completion, an average of 3 year
  The change between baseline A-DQOL score and A-DQOL score 3 years after admission. CA-DQOL has maximum score of 230. Subscale 1 measures life satisfaction and has 15 questions, each question has a minimum score of 1 (indicates very unsatisfied), maximum score of 5(indicates very satisfied). Subscale 2 measures frequency of diabetes affects life quality, has 20 questions, each question has a minimum score of 1 (indicates never affect life quality), maximum score of 5(indicates always affect life quality). Subscale 3 measures how much the patient worries about how diabetes affects daily life and has 7 questions, each question has a minimum score of 1 (indicates never worries), maximum score of 5(indicates very worries). Subscale 4 measures how much the patient worries about the diabetes-related conditions and has 4 questions, each question has a minimum score of 1 (indicates never worries), maximum score of 5(indicates very worries).
Morisky scale score change | through study completion, an average of 3 year
  The change between baseline Morisky score and Morisky score 3 years after admission. Morisky scale measures patients' compliance of medication usage. The Morisky scale has 4 questions, each question has a minimum score of 0 (did not comply the medical instruction), maximum score of 1(comply medical instruction). the scale has totally 4 scores
DASS-C21scale score change | through study completion, an average of 3 year
  The change between baseline DASS-C21 scale score and DASS-C21 scale score 3 years after admission. DASS-C21 scale is Depression Anxiety Stress Scale 21 scale in Chinese. The scale measures patients' level of depression, anxiety and stress. The scale has 21 questions, each question has a minimum score of 0 (did not meet the description), maximum score of 3(completely meet the description). the scale has totally 63 scores

OTHER OUTCOMES:
Diabetes complications | through study completion, an average of 3 year
  Newly diagnosed diabetes complications (Diabetic nephropathy, diabetic retinopathy, diabetic neuropathy, diabetic lower extremity arterial disease, diabetic foot)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] International Diabetes Federation. IDF Diabetes Atlas. Brussels, Belgium: International Diabetes Federation 8th edition; 2017
- [Background] [A mass survey of diabetes mellitus in a population of 300,000 in 14 provinces and municipalities in China (author's transl)]. Zhonghua Nei Ke Za Zhi. 1981 Nov;20(11):678-83. No abstract available. Chinese. PMID 7341098
- [Background] Pan XR, Yang WY, Li GW, Liu J. Prevalence of diabetes and its risk factors in China, 1994. National Diabetes Prevention and Control Cooperative Group. Diabetes Care. 1997 Nov;20(11):1664-9. doi: 10.2337/diacare.20.11.1664. PMID 9353605
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Wang L, Gao P, Zhang M, Huang Z, Zhang D, Deng Q, Li Y, Zhao Z, Qin X, Jin D, Zhou M, Tang X, Hu Y, Wang L. Prevalence and Ethnic Pattern of Diabetes and Prediabetes in China in 2013. JAMA. 2017 Jun 27;317(24):2515-2523. doi: 10.1001/jama.2017.7596. PMID 28655017
- [Background] Ji LN, Lu JM, Guo XH, Yang WY, Weng JP, Jia WP, Zou DJ, Zhou ZG, Yu DM, Liu J, Shan ZY, Yang YZ, Hu RM, Zhu DL, Yang LY, Chen L, Zhao ZG, Li QF, Tian HM, Ji QH, Liu J, Ge JP, Shi LX, Xu YC. Glycemic control among patients in China with type 2 diabetes mellitus receiving oral drugs or injectables. BMC Public Health. 2013 Jun 21;13:602. doi: 10.1186/1471-2458-13-602. PMID 23800082
- [Background] Wan EYF, Fung CSC, Jiao FF, Yu EYT, Chin WY, Fong DYT, Wong CKH, Chan AKC, Chan KHY, Kwok RLP, Lam CLK. Five-Year Effectiveness of the Multidisciplinary Risk Assessment and Management Programme-Diabetes Mellitus (RAMP-DM) on Diabetes-Related Complications and Health Service Uses-A Population-Based and Propensity-Matched Cohort Study. Diabetes Care. 2018 Jan;41(1):49-59. doi: 10.2337/dc17-0426. Epub 2017 Nov 14. PMID 29138274
- [Background] American Diabetes Association. (11) Children and adolescents. Diabetes Care. 2015 Jan;38 Suppl:S70-6. doi: 10.2337/dc15-S014. No abstract available. PMID 25537712
- [Background] Type 2 diabetes in adults: management. London: National Institute for Health and Care Excellence (NICE); 2015 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK338142/ PMID 26741015
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Wagner EH, Grothaus LC, Sandhu N, Galvin MS, McGregor M, Artz K, Coleman EA. Chronic care clinics for diabetes in primary care: a system-wide randomized trial. Diabetes Care. 2001 Apr;24(4):695-700. doi: 10.2337/diacare.24.4.695. PMID 11315833